CLINICAL TRIAL: NCT01301066
Title: A 12-Week, Randomized, Double-Blind, Active-Controlled, Parallel-Group Study Comparing Pitavastatin 4 mg vs. Pravastatin 40 mg in HIV-Infected Subjects With Dyslipidemia, Followed by a 40-Week Safety Extension Study
Brief Title: A 12-Week Study Comparing Pitavastatin 4 mg vs. Pravastatin 40 mg in HIV-Infected Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Collaborators: Kowa Pharmaceuticals America, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NK-104-4.05US
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — pitavastatin; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin 4 mg QD (Experimental)
  Interventions: Drug: Pitavastatin
- Pravastatin 40 mg QD (Active Comparator)
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 4 mg QD
  Other Names: Livalo
  Arms: Pitavastatin 4 mg QD
Drug: Pravastatin — Pravastatin 40 mg QD
  Arms: Pravastatin 40 mg QD

SUMMARY:
A 12-Week, Randomized, Double-Blind, Active-Controlled, Parallel-Group Study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (non-pregnant, non-lactating females) 18-70 years of age, inclusive, at time of consent.
* Both men and women of child bearing potential (i.e., not surgically sterile or post-menopausal defined as age >40 years without menses for ≥2 years) must agree to use at least 2 reliable forms of contraception
* Documented HIV infection.

Exclusion Criteria:

* Homozygous familial hypercholesterolemia
* Any conditions that may cause secondary dyslipidemia
* History of coronary artery disease (CAD) or CAD equivalent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Costa Mesa, California
  - Long Beach, California
  - Los Angeles, California
  - Newport Beach, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Coral Gables, Florida
  - Fort Lauderdale, Florida
  - Ft. Pierce, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Springfield, Massachusetts
  - Berkley, Michigan
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - Randolph Township, New Jersey
  - New York, New York
  - Rochester, New York
  - Huntersville, North Carolina
  - Addison, Texas
  - Austin, Texas
  - Corpus Christi, Texas
  - Fort Worth, Texas
  - Harlingen, Texas
  - Houston, Texas
  - Longview, Texas
  - Annandale, Virginia
  - Seattle, Washington
  - Spokane, Washington

REFERENCES:
- [Derived] Aberg JA, Sponseller CA, Ward DJ, Kryzhanovski VA, Campbell SE, Thompson MA. Pitavastatin versus pravastatin in adults with HIV-1 infection and dyslipidaemia (INTREPID): 12 week and 52 week results of a phase 4, multicentre, randomised, double-blind, superiority trial. Lancet HIV. 2017 Jul;4(7):e284-e294. doi: 10.1016/S2352-3018(17)30075-9. Epub 2017 Apr 13. PMID 28416195
- [Derived] Toribio M, Fitch KV, Sanchez L, Burdo TH, Williams KC, Sponseller CA, McCurdy Pate M, Aberg JA, Zanni MV, Grinspoon SK. Effects of pitavastatin and pravastatin on markers of immune activation and arterial inflammation in HIV. AIDS. 2017 Mar 27;31(6):797-806. doi: 10.1097/QAD.0000000000001427. PMID 28252528
- [Derived] Joshi PH, Miller PE, Martin SS, Jones SR, Massaro JM, D'Agostino RB Sr, Kulkarni KR, Sponseller C, Toth PP. Greater remnant lipoprotein cholesterol reduction with pitavastatin compared with pravastatin in HIV-infected patients. AIDS. 2017 Apr 24;31(7):965-971. doi: 10.1097/QAD.0000000000001423. PMID 28121706

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pitavastatin 4 mg QD | Pravastatin 40 mg QD
Started | 126 | 126
Completed | 99 | 91
Not Completed | 27 | 35
Not completed — Lost to Follow-up | 5 | 11
Not completed — Protocol Violation | 8 | 7
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Adverse Event | 6 | 6
Not completed — Sponsor Decision | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 4 mg QD | Pravastatin 40 mg QD | Total
Number analyzed (Participants) | 126 | 126 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 126 | 252
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 106 | 111 | 217
Region of Enrollment [Number; unit: participants]
  United States | 126 | 126 | 252

OUTCOME MEASURES:

1. Primary Outcome: Change of Fasting Serum Low-density Lipoprotein Cholesterol (LDL-C) at 12 Weeks
Time Frame: 12 weeks minus baseline
Population: modified Intent To Treat (mITT) population included all randomized subjects who received at least 1 dose of study drug and had at least 1 on-treatment lipid assessment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pitavastatin 4 mg QD | Pravastatin 40 mg QD
Number analyzed (Participants) | 121 | 126
mg/dL | 155.1 (25.93) | 154.6 (23.91)

ADVERSE EVENTS:
Arm/Group | Pitavastatin 4 mg QD | Pravastatin 40 mg QD
Serious Adverse Events (participants affected / at risk) | 7/126 | 3/126
Other Adverse Events (participants affected / at risk) | 10/126 | 5/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pitavastatin 4 mg QD (N=126) | Pravastatin 40 mg QD (N=126)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial septal defect (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Herpes dermatitis (Infections and infestations) | 1 (1) | 0 (0)
Multiple fractures (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.6% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4 mg QD (N=126) | Pravastatin 40 mg QD (N=126)
Fatigue (General disorders) | 2 | 1
Headache (General disorders) | 2 | 1
Upper abdominal pain (Gastrointestinal disorders) | 2 | 0
Blood CK increased (Blood and lymphatic system disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have the right to the first publication of the results of the Study. PI may publish, however PI must submit publication to sponsor for review at least 60 days prior to proposed publication. Sponsor may remove any information that is considered confidential and/or proprietary.